CLINICAL TRIAL: NCT02235649
Title: Exploring the Feasibility of Social Skills Training in People With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychiatry, London (Other)
Responsible Party: Principal Investigator, Matteo Cella, Lecturer in Clinical Psychology, Institute of Psychiatry, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13/LO/1791
Record Dates: First submitted 2014-04-01; First posted 2014-09-10 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Focus of Study

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAU (No Intervention): Treatment as usual
- SOC+TAU (Active Comparator): Social Cognition intervention + Treatment as Usual
  Interventions: Behavioral: Social Cognition therapy ( Psychological Therapy)

INTERVENTIONS:
Behavioral: Social Cognition therapy ( Psychological Therapy)
  Arms: SOC+TAU

SUMMARY:
Reduced social and community functioning is a predominant and enduring feature in people experiencing severe mental illness such as psychosis. The large majority of interventions (mostly pharmacological) target the so called positive symptoms (e.g. hallucinations and delusions) but poorly address functional and social consequences of the illness.

This study attempts to fill this gap by assessing the feasibility and acceptability of a psychological intervention targeting social cognition deficit in people with psychosis. The intervention is a group psychological treatment facilitated by a clinical psychologist targeting competencies such as emotion recognition, social situation appraisal and guessing people's intentions and mental states. The group therapy takes advantage of audiovisual material to illustrate strategies and thinking styles that may help participants to overcome difficulties in social settings.

A second objective of this study is to test a new method to measure social cognition. Recent research showed that interview and performance based tests are poorly associated with every day activity of people with schizophrenia. This study is planning to evaluate the feasibility of new assessment methods for social cognition in everyday life using portable electronic devices (Experience Sampling Method and an activity watch). These devices will be carried by participants in their everyday life and will ask about feelings and levels of social activities at random times and record basic physiological and activity levels.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis part of the psychosis spectrum (according to DSM-IV or DSM-V or ICD-10); age 18-65 yrs; good command of the English language; social engagement problems as evidenced by care coordinator report and number of hours spent in social activities per week lower than 10.

Exclusion Criteria:

Primary diagnosis of substance abuse disorder; change in antipsychotic medication in the last six weeks; significant learning difficulties (premorbid IQ lower than 70).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability | 10 weeks
  Number of sessions attended and number of drop out from therapy. Acceptability is assesses with a questionnaire designed for psychological interventions (Gledhill et al., 1998).

SECONDARY OUTCOMES:
Effectiveness (i.e. social behaviour and social cognition) | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, King's College London, London, United Kingdom